CLINICAL TRIAL: NCT07346690
Title: Acute Dose-Dependent Effects of Oral THC on Physiological and Subjective Responses in Healthy Cannabis-Experienced Adults
Brief Title: A Study Testing the Effects of Different THC Doses on Psychological and Biological Function
Acronym: DRATT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DRATT
Record Dates: First submitted 2025-12-16; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Evaluate PK Profile; Evaluate PD Profile; Healthy Adults; Safety and Tolerability in Healthy Volunteers
Keywords: Cannabinoid; Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral Study Drug: AVCN6mg -> AVCN9mg -> AVCN15mg -> Placebo (Experimental): 3 Doses of AVCN319301b (6mg, 9mg, 15mg) and placebo, each separated by >1 week washout period. Each participant receives all interventions in a double-blind randomized order based on a 4 sequence reverse Williams crossover design.
  Interventions: Drug: AVCN319301b (6mg); Drug: AVCN319301b (9mg); Drug: AVCN319301b (15mg); Drug: Placebo
- Oral Study Drug: AVCN9mg -> AVCN15mg -> Placebo -> AVCN6mg (Experimental): 3 Doses of AVCN319301b (6mg, 9mg, 15mg) and placebo, each separated by >1 week washout period. Each participant receives all interventions in a double-blind randomized order based on a 4 sequence reverse Williams crossover design.
  Interventions: Drug: AVCN319301b (6mg); Drug: AVCN319301b (9mg); Drug: AVCN319301b (15mg); Drug: Placebo
- Oral Study Drug: AVCN15mg -> Placebo -> AVCN6mg -> AVCN9mg (Experimental): 3 Doses of AVCN319301b (6mg, 9mg, 15mg) and placebo, each separated by >1 week washout period. Each participant receives all interventions in a double-blind randomized order based on a 4 sequence reverse Williams crossover design.
  Interventions: Drug: AVCN319301b (6mg); Drug: AVCN319301b (9mg); Drug: AVCN319301b (15mg); Drug: Placebo
- Oral Study Drug: Placebo -> AVCN6mg -> AVCN9mg -> AVCN15mg (Experimental): 3 Doses of AVCN319301b (6mg, 9mg, 15mg) and placebo, each separated by >1 week washout period. Each participant receives all interventions in a double-blind randomized order based on a 4 sequence reverse Williams crossover design.
  Interventions: Drug: AVCN319301b (6mg); Drug: AVCN319301b (9mg); Drug: AVCN319301b (15mg); Drug: Placebo

INTERVENTIONS:
Drug: AVCN319301b (6mg) — AVCN319301b is a standardized oral capsule containing a precise dose of Δ9-THC.
  Other Names: Low Dose
Drug: AVCN319301b (9mg) — AVCN319301b is a standardized oral capsule containing a precise dose of Δ9-THC.
  Other Names: Medium Dose
Drug: AVCN319301b (15mg) — AVCN319301b is a standardized oral capsule containing a precise dose of Δ9-THC.
  Other Names: High Dose
Drug: Placebo — The matched placebo is an oral capsule identical in appearance to the active study drug and contains the same non-medicinal ingredients but no Δ9-THC. It is manufactured to match the active capsules in size, color, taste, and packaging to maintain blinding for participants and study staff.

SUMMARY:
The goal of this clinical trial is to learn how a investigational medicinal product (THC) affects psychological and physical responses in healthy adults with prior cannabis use experience. The main questions it aims to answer are:

- How do different dose levels of the investigational medicinal product (THC) influence short-term subjective and physiological responses?

Researchers will compare three dose levels of the study drug to a placebo (a look-alike substance with no active ingredient) to see how responses vary across sessions.

Participants will:

* Attend four in-person study visits, each involving a single dose of either the study drug or placebo
* Complete questionnaires about their moment-to-moment experiences
* Have their heart rate, blood pressure, and other physical measures monitored
* Undergo serial blood sampling to measure circulating biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55
* No major medical or psychiatric conditions
* At least one previous, well-tolerated experience with cannabis
* Not currently pregnant or breastfeeding

Exclusion Criteria:

* Family history (first- or second-degree relatives) of bipolar disorder, psychosis, or schizophrenia
* Significant negative reaction to cannabis in the past or known allergy to cannabis products
* Currently using recreational drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory - State | Baseline and multiple points up to 300 minutes post-dose.
  The STAI-S is a validated self-report questionnaire that measures how anxious or calm a person feels "right now." Participants rate statements about current stress, worry, or relaxation on a 4-point scale. Scores are summed to provide a total anxiety rating. Higher scores reflect greater momentary anxiety. This measure is repeated throughout each session to track short-term changes in emotional state following study drug or placebo.

SECONDARY OUTCOMES:
Subjective Drug Effects (Drug Effects Questionnaire; DEQ) | Baseline and multiple points up to 300 minutes post-dose.
  The DEQ is a brief self-report scale assessing immediate subjective reactions to the study drug. Participants rate sensations such as "feel drug effects," "feel high," or "like the drug" on visual analog scales. This measure captures moment-to-moment changes in subjective experience across the session.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Adverse event recording begins with receiving the first dose of investigational medicinal product and ends one week following the last dose of investigational medicinal product (end of study).
  All adverse events reported by participants or observed by study staff are recorded and categorized by severity and relatedness to the investigational medicinal product
Mood States (Profile of Mood States; POMS) | Baseline and multiple points up to 300 minutes post-dose.
  The POMS measures transient emotional states such as tension, calmness, fatigue, and well-being. Participants rate how they feel using a list of adjectives. Scores reflect current mood and allow researchers to track short-lived emotional changes across the study period.
Positive and Negative Affect (PANAS-SF) | Baseline and multiple points up to 300 minutes post-dose.
  The PANAS-SF asks participants to rate the extent to which they feel various positive and negative emotions. Scores give a snapshot of emotional tone during the session.
Heart Rate | Continuous measurements from baseline to 300 minutes post-dose.
  Heart rate is measured using an automated vital-signs monitor while the participant is seated.
Heart Rate Variability | Continuous measurements from baseline to 300 minutes post-dose.
  Heart Rate Variability represents natural variation in the time between heartbeats and is calculated from continuous pulse or ECG-based data.
  - Systolic and diastolic blood pressure are obtained with an automated cuff.
Blood Pressure | Continuous measurements from baseline to 300 minutes post-dose.
  Systolic and diastolic blood pressure are obtained with an automated cuff.
Cortisol Levels | Blood samples collected at multiple points from baseline to 300 minutes post-dose.
  Cortisol is a hormone released during stress. Plasma cortisol concentrations are measured from venous blood samples using laboratory assays.
Endocannabinoid Levels | Blood samples collected at multiple points from baseline to 300 minutes post-dose.
  Endocannabinoids (AEA, 2-AG, PEA, OEA) and related lipids are naturally occurring signaling molecules. Plasma endocannabinoids are measured from venous blood samples using specialized laboratory techniques (e.g., LC-MS/MS).
Cmax of Δ9-THC and its Metabolites | Blood samples collected at multiple points from baseline to 300 minutes post-dose.
  Plasma Δ9-THC and its Metabolites (THC, 11-OH-THC, THC-COOH) are measured from venous blood samples using specialized laboratory techniques (e.g., LC-MS/MS) to calculate Cmax.
Tmax of Δ9-THC and its Metabolites | Blood samples collected at multiple points from baseline to 300 minutes post-dose.
  Plasma Δ9-THC and its Metabolites (THC, 11-OH-THC, THC-COOH) are measured from venous blood samples using specialized laboratory techniques (e.g., LC-MS/MS) to calculate Tmax.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Heritage Medical Research Building, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided